CLINICAL TRIAL: NCT01232413
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Active-Controlled Crossover Study to Evaluate the Effect of Repeat Oral Doses of ASP1941 on Cardiac Repolarization in Healthy Male and Female Adult Subjects
Brief Title: A Study of the Effect of ASP1941 on Cardiac Repolarization in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 1941-CL-0058
Record Dates: First submitted 2010-10-27; First posted 2010-11-02 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Cardiac Repolarization
Keywords: Thorough QT (TQT); ASP1941
MeSH Terms: interventions — ipragliflozin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Treatment B (Experimental): ASP1941 low dose
  Interventions: Drug: ASP1941
- Treatment C (Experimental): ASP1941 high dose
  Interventions: Drug: ASP1941
- Treatment D (Active Comparator): Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Placebo — Oral
  Arms: Treatment A
Drug: ASP1941 — Oral
  Arms: Treatment B; Treatment C
Drug: Moxifloxacin — Oral
  Other Names: Avelox
  Arms: Treatment D

SUMMARY:
The objective of this study is to evaluate the effect of repeat oral dosing of ASP1941 on electrocardiogram (ECG) measurements.

DETAILED DESCRIPTION:
Subjects will be randomized in four treatment sequences of twenty subjects each. Subjects in each treatment sequence will participate in a total of four treatment periods (A, B, C, and D) separated by washout periods of at least 7 days from completion of the prior period (Day 8) through clinical check-in (Day -1) of the next study period.

For Period 1, subjects will be admitted to the clinical research unit on Day -2. For each subsequent study period, subjects will be admitted to the clinical research unit on Day -1. Subjects will be discharged from the unit after completing procedures on Day 8 of each period. Subjects will receive a follow-up telephone call 7-10 days after their last clinic day (Period 4\Early Discontinuation [ED]).

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 45 kg, and has a body mass index (BMI) of 18 to 32 kg/m2
* If female, subject must be at least two years postmenopausal, surgically sterile or practicing effective birth control, and not pregnant or lactating
* The male or female subject agrees to practice highly effective birth control until 30 days post last study drug dose
* The subject is highly likely to comply with the protocol-defined procedures and complete the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death due to cardiac causes at a young age of a close relative)
* The subject anticipates an inability to abstain from alcohol, or caffeine use, or from grapefruit and grapefruit juice from 72 hours prior to dosing and throughout the duration of the study
* The subject has used tobacco-containing products and nicotine or nicotine-containing products within past six months
* The subject is unable to tolerate a controlled, quiet study conduct environment, including avoidance during specified times (e.g., prior to and in ECG extraction windows) of music, TV, movies, games and activities that may cause excitement, emotional tension or arousal
* The subject is unwilling to comply with study rules, including attempting to void at specified times (e.g., prior to ECG extraction windows), remaining quiet, awake, undistracted, motionless and supine during specified times, and avoiding vigorous exercise as directed
* The subject is unable to tolerate study-specific diet
* The subject has a history or evidence of any clinically significant cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy (excluding non-melanoma skin cancer)
* The subject has a history of clinically significant allergic conditions or anaphylactic reactions
* The subject has any condition possibly affecting drug absorption
* The subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous)infection within 1 week prior to clinic check in for any treatment period
* The subject is known positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive test for hepatitis C antibody, or positive for hepatitis B antigen (HBsAg)
* The subject has used prescription or non-prescription drugs within 14 days or 5-half lives (whichever is longer) or complementary and alternative medicines (CAM) within 28 days prior to Day -2 of Period 1 (excluding oral contraceptives, hormone replacement therapy [HRT], and acetaminophen)
* The subject has received an experimental agent within 30 days or 10 half-lives, whichever is longer, prior to study drug administration
* The subject is participating in another clinical trial or has participated in another dose group of the current trial
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
QTcF evaluated through electrocardiogram analysis (ECG) | Days -1, 1 and 7 (period 1) and Days 1 and 7 (period 2-4)
  QTcF is a QT interval corrected for heart rate (Fridericia's formula)

SECONDARY OUTCOMES:
Evaluation of Electrocardiogram (ECG) | Days -1, 1 and 7 (period 1) and Days 1 and 7 (period 2-4)
QTcI evaluated through electrocardiogram analysis | Days -1, 1 and 7 (period 1) and Days 1 and 7 (period 2-4)
  QTcI is a QT interval corrected for individual heart rate
QTcB evaluated through electrocardiogram analysis (ECG) | Days -1, 1 and 7 (period 1) and Days 1 and 7 (period 2-4)
  QTcB is a QT interval corrected for heart rate (Bazett's formula)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- West Bend, Wisconsin, United States

REFERENCES:
- [Derived] Zhang W, Smulders R, Abeyratne A, Dietz A, Krauwinkel W, Kadokura T, Keirns J. Ipragliflozin does not prolong QTc interval in healthy male and female subjects: a phase I study. Clin Ther. 2013 Aug;35(8):1150-1161.e3. doi: 10.1016/j.clinthera.2013.06.009. Epub 2013 Aug 2. PMID 23910665